CLINICAL TRIAL: NCT02641730
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo Controlled Study Evaluating the Efficacy and Safety of Guselkumab for the Treatment of Subjects With Palmoplantar Pustulosis
Brief Title: An Efficacy and Safety of Guselkumab in Participants With Palmoplantar Pustulosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108046; CNTO1959PPP3001 (Other: Janssen Pharmaceutical K.K.)
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Palmoplantar Pustulosis
Keywords: Guselkumab; CNTO 1959; Placebo; Palmoplantar Pustulosis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive guselkumab 200 milligram (mg) at Week 0, 4, 12 and every 8 weeks thereafter through Week 60, and two syringes of placebo at Week 16 to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2 (Experimental): Participants will receive a syringe of guselkumab 100 mg and a syringe of placebo for guselkumab at Week 0, 4, 12 and every 8 weeks thereafter through Week 60, two syringes of placebo at Week 16 to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 3 (Experimental): Participants will receive two syringes of placebo at Week 0, 4 and 12. At Week 16, placebo participants will be randomized in a 1:1 ratio to guselkumab mg arm (Group 3a) or 100 mg arm (Group 3b). Group 3a participants will receive guselkumab 200 mg at Week 16, 20 and every 8 weeks thereafter through Week 60. Group 3b participants will receive guselkumab 100 mg and a syringe of placebo at Week 16, 20 and every 8 weeks thereafter through Week 60.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive two or one syringe of guselkumab 100 mg subcutaneously at Week 0, 4, 12 and every 8 weeks thereafter through Week 60 in group 1 or 2. Group 3a or 3b participants will receive two or one syringe of guselkumab 100 mg at Week 16, 20 and every 8 weeks thereafter through Week 60.
  Other Names: CNTO 1959
Drug: Placebo — Participants in group 1 will receive placebo at Week 16. Participants in group 2 will receive placebo at Week 0, 4, 12, 16, 20 and every 8 weeks thereafter through Week 60. Participants in group 3 will receive placebo at Week 0, 4, 12, then at Week 16, 20 and every 8 weeks thereafter through Week 60 for group 3b.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of guselkumab for the treatment of participants with palmoplantar pustulosis.

DETAILED DESCRIPTION:
This is a phase 3, randomized (study drug assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), multicenter (when more than one hospital works on a medical research study) placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study) study in participants with palmoplantar pustulosis. The study will consist of 3 phases: screening phase (up to 6 weeks), treatment period (week 0 - week 60) and observational period (up to week 84). Participants will be assigned to 1 of 3 treatment groups (200 milligram [mg] guselkumab, 100 mg guselkumab or placebo group) using a stratified block randomization method in a 1:1:1 ratio at Week 0 and Group III (placebo) participants will be allocated in a 1:1 ratio to 1 of 2 treatment groups at Week 16. Participants will primarily be assessed for change from baseline in Palmo-Plantar Pustular Area and Severity Index (PPPASI) total score at Week 16. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of palmoplantar pustulosis (with or without pustulotic arthro-osteitis, concurrent extra-palmoplantar lesions) for at least 24 weeks before screening
* Has a >= 12 PPPASI total score at screening and at baseline
* Has a moderate or more severe pustules/vesicle on the palms or soles (>= 2 PPPASI severity score) at screening and baseline
* Has inadequate response to the treatment with topical steroid and/or topical vitamin D3 derivative preparations and/or the phototherapy and/or systemic etretinate prior to or at screening. Inadequate response is defined as a case judged by the investigator
* Before the first administration of study drug, a woman must be either: Not of childbearing potential: premenarchal; postmenopausal or Of childbearing potential and practicing a highly effective method of birth control

Exclusion Criteria:

* Has a diagnosis of plaque-type psoriasis
* Has obvious improvement during screening (>= 5 PPPASI total score improvement during the screening)
* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has unstable cardiovascular disease, defined as a recent clinical deterioration (eg, unstable angina, rapid atrial fibrillation) in the last 12 weeks or a cardiac hospitalization within the last 12 weeks before screening
* Currently has a malignancy or has a history of malignancy within 5 years before screening (with the exception of a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 12 weeks before screening or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 12 weeks before screening)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (32):
- Japan (32):
  - Asahikawa
  - Fukuoka
  - Fukushima
  - Hachiōji
  - Hokkaido
  - Ichikawa
  - Ichinomiya
  - Kahoku-District
  - Kanazawa
  - Kobe
  - Kochi
  - Kofu
  - Kumamoto
  - Kyoto
  - Matsumoto
  - Morioka
  - Nagasaki
  - Nagoya
  - Osaka
  - Ōsaka-sayama
  - Sagamihara
  - Saku
  - Shimotsuke
  - Suita-shi
  - Takamatsu
  - Tokushima
  - Tokyo
  - Toyoake
  - Tōon
  - Tsu
  - Tsukuba
  - Yokohama

REFERENCES:
- [Derived] Terui T, Kobayashi S, Okubo Y, Murakami M, Zheng R, Morishima H, Goto R, Kimura T. Efficacy and Safety of Guselkumab in Japanese Patients With Palmoplantar Pustulosis: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2019 Oct 1;155(10):1153-1161. doi: 10.1001/jamadermatol.2019.1394. PMID 31268476

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to guselkumab subcutaneous (SC) injection at Weeks 0, 4, and 12 during placebo-controlled period (PCP). At Week 16 placebo participants were randomized to receive guselkumab 200 milligram (mg) or 100 mg.
- Placebo Then Guselkumab 100 mg: Participants who received placebo matched to guselkumab SC injection through Week 16 during placebo-controlled period were crossed over to receive guselkumab 100 mg SC injection at Week 16 and 20 and every 8 Weeks thereafter through Week 60. All participants who continued the study at Week 60 in this group were observed until Week 84 without receiving the study drug.
- Placebo Then Guselkumab 200 mg: Participants who received placebo matched to guselkumab SC injection through Week 16 during placebo-controlled period were crossed over to receive guselkumab 200 mg SC injection at Week 16 and 20 and every 8 Weeks thereafter through Week 60. All participants who continued the study at Week 60 in this group were observed until Week 84 without receiving the study drug.
- Guselkumab 100 mg: Participants received guselkumab 100 mg SC injection at Weeks 0, 4, and 12 and once every 8 Weeks thereafter through Week 60 and placebo matched to guselkumab SC injection at Week 16 to maintain the blind. All participants who continued the study at Week 60 in this group were observed from until Week 84 without receiving the study drug.
- Guselkumab 200 mg: Participants received guselkumab 200 mg SC injection at Weeks 0, 4, and 12 and thereafter once every 8 Weeks through Week 60 and placebo matched to guselkumab SC injection at Week 16 to maintain the blind. All participants who continued the study at Week 60 in this group were observed until Week 84 without receiving the study drug.
Period: Placebo Controlled Period (Week 0 - 16)
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Started | 53 | 0 | 0 | 54 | 52
Completed | 51 | 0 | 0 | 53 | 50
Not Completed | 2 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 2
Period: After Controlled Period (Week 16 - 52)
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Started | 0 | 25 | 26 | 53 | 50
Completed | 0 | 21 | 24 | 45 | 44
Not Completed | 0 | 4 | 2 | 8 | 6
Not completed — Adverse Event | 0 | 1 | 1 | 5 | 4
Not completed — Lack of Efficacy | 0 | 2 | 0 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 1 | 1 | 0 | 1
Period: Observational Period (Week 60 - Week 84)
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Started | 0 | 21 | 24 | 45 | 44
Completed | 0 | 21 | 24 | 45 | 43
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab 100 mg | Guselkumab 200 mg | Total
Number analyzed (Participants) | 53 | 54 | 52 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (8.14) | 53.9 (10.88) | 52.9 (13.39) | 53.3 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 36 | 126
  Male | 9 | 8 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 53 | 54 | 52 | 159
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 53 | 54 | 52 | 159
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 53 | 54 | 52 | 159

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Palmoplantar Pustulosis Area and Severity Index (PPPASI) Total Score at Week 16
Description: PPPASI assesses severity of palmoplantar pustulosis (PPP) lesions and response to therapy. In PPPASI, palms, soles are divided into 4 regions: right palm(RP), left palm(LP), right sole(RS), left sole(LS), that account for 20 percent (%), 20%,30%,30%, respectively, of total surface area(TSA) of palms, soles. Each area is assessed separately for erythema(E), pustules/vesicles (P), desquamation/scales (D), each rated on a scale (0-4). PPPASI produces score range of 0-72 using formula, PPPASI=(E+P+D)Area*0.2(RP)+(E+P+D)Area*0.2 (LP)+(E+P+D)Area*0.3(RS)+(E+P+D)Area*0.3(LS). Higher a score more the severe disease. Participants who discontinue study agent as they met treatment failure(TF) criterion(lack of efficacy/AE of worsening of PPP/who started a protocol-prohibited medication/therapy that could improve PPP), their baseline value carried forward to post baseline attending visits before and at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Baseline and Week 16
Population: Randomized analysis set: all randomized participants at Week 0, whether they received study treatment or not and had any post-baseline efficacy assessment. Missing values were imputed based on TF criterion, last observation carried forward (LOCF) method till Week 60;no imputation performed for missing data after Week 60 (in observational period).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 54 | 52
Units on a scale | -7.79 (10.596) | -15.08 (11.252) | -11.07 (7.779)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg; Test type: Superiority; p < 0.001, Mixed-Model for Repeated Measures; Mean Difference (Final Values) = -7.69, 95% CI 2-sided [-11.000 to -4.383], Standard Error of Mean 1.674
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 200 mg; Test type: Superiority; p = 0.017, Mixed-Model for Repeated Measures; Mean Difference (Final Values) = -4.11, 95% CI 2-sided [-7.468 to -0.748], Standard Error of Mean 1.700

2. Secondary Outcome: Change From Baseline in Palmoplantar Severity Index (PPSI) Total Score at Week 16
Description: PPSI assesses the severity of PPP lesions and their response to therapy with a score ranging from 0 to 12. A higher score indicates more severe disease. In the PPSI system, the more severely affected location (palms or soles) were to be identified as the evaluation sites at screening that to be assessed at all subsequent visits. Evaluation sites were assessed separately for erythema, pustules/vesicles and desquamation/scale, for most severe skin lesion rated on a scale of 0 to 4. Participants who discontinue study agent as they met a TF criterion, their baseline value carried forward to the post-baseline attending visits before and at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Baseline and Week 16
Population: Population included Randomized analysis set. The missing values were imputed based on Treatment Failure (TF) criterion and last scheduled observation carried forward (LOCF) method until Week 60; no imputation performed for missing data after Week 60 (in observational period).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 54 | 52
Units on a scale | -2.0 (2.41) | -3.9 (2.94) | -3.0 (2.57)

3. Secondary Outcome: Percentage of Participants Who Achieved a PPPASI-50 Response at Week 16
Description: PPPASI assesses severity of PPP lesions and their response to therapy. In PPPASI system, palms and soles are divided into 4 regions: right palm, left palm, right sole, and left sole, that account for 20%, 20%, 30%, and 30%, respectively, of TSA of palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicles, and desquamation/scales, each rated on a scale of 0 to 4. PPPASI produces a score range from 0 to 72. Higher score indicates more severe disease. PPPASI-50 response represents participants who achieved at least a 50% improvement from baseline in the PPPASI score. Participants who discontinue study agent as they met a TF criterion were considered as non-responders at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 16
Population: Population included Randomized analysis set. The missing values were imputed based on TF criterion and LOCF method until Week 60; no imputation performed for missing data after Week 60 (in observational period).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 54 | 52
Percentage of participants | 34.0 | 57.4 | 36.5

4. Secondary Outcome: Change From Baseline in PPPASI Total Score
Description: PPPASI assesses severity of PPP lesions and their response to therapy. In PPPASI system, palms and soles are divided into 4 regions: right palm, left palm, right sole, and left sole, which account for 20%, 20%, 30%, and 30%, respectively, of TSA of palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicles, and desquamation/scales, each rated on a scale of 0 to 4. PPPASI produces a score range from 0 to 72. Higher score indicates more severe disease. PPPASI-50 response represents participants who achieved at least a 50% improvement from baseline in the PPPASI score. Participants were analyzed according to the treatment at Week 0 or 16. Participants who discontinue study agent as they met a TF criterion, their baseline value carried forward to the post-baseline attending visits before and at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Baseline, Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: Population included Randomized analysis set. The missing values were imputed based on TF criterion and LOCF method until Week 60; no imputation performed for missing data after Week 60 (in observational period). Here 'n' signifies the number of participants analyzed at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Units on a scale
  Change at week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 2 | -3.58 (5.303) |  |  | -2.27 (6.832) | -3.02 (5.829)
  Change at week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 4 | -4.39 (6.805) |  |  | -6.43 (7.907) | -5.28 (5.692)
  Change at week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 8 | -6.31 (7.986) |  |  | -10.60 (8.358) | -7.94 (7.305)
  Change at week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 12 | -7.60 (9.197) |  |  | -12.80 (9.706) | -9.35 (8.121)
  Change at week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 20 |  | -12.33 (9.672) | -8.66 (11.032) | -16.33 (11.350) | -13.76 (8.278)
  Change at week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 24 |  | -14.45 (9.878) | -10.90 (10.759) | -17.86 (11.219) | -15.38 (8.864)
  Change at week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 28 |  | -15.44 (10.597) | -13.90 (11.383) | -18.32 (11.425) | -16.86 (9.443)
  Change at week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 32 |  | -16.92 (10.615) | -15.63 (10.789) | -18.52 (11.544) | -17.64 (9.792)
  Change at week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 36 |  | -18.15 (11.372) | -17.19 (11.199) | -18.87 (11.909) | -17.72 (10.083)
  Change at week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 40 |  | -19.06 (11.683) | -18.63 (10.812) | -18.85 (12.356) | -18.54 (9.887)
  Change at week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 44 |  | -18.92 (12.099) | -18.77 (11.119) | -18.91 (12.338) | -18.61 (10.093)
  Change at week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 48 |  | -19.54 (12.572) | -19.18 (10.547) | -19.72 (12.506) | -18.99 (9.686)
  Change at week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 52 |  | -20.04 (12.362) | -18.88 (11.635) | -19.95 (12.567) | -19.63 (9.776)
  Change at week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 60 |  | -20.18 (11.880) | -19.62 (11.566) | -20.17 (12.829) | -20.37 (10.098)
  Change at week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Change at week 72 |  | -22.09 (11.958) | -21.08 (11.855) | -22.13 (10.400) | -22.05 (9.136)
  Change at week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Change at week 84 |  | -22.60 (11.781) | -21.19 (13.619) | -21.32 (10.458) | -22.56 (9.352)

5. Secondary Outcome: Change From Baseline in PPSI Total Score
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Units on a scale
  Change at week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 2 | -0.5 (1.14) |  |  | -0.5 (1.68) | -0.6 (1.35)
  Change at week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 4 | -0.7 (1.26) |  |  | -1.5 (2.14) | -1.3 (1.94)
  Change at week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 8 | -1.2 (1.70) |  |  | -2.6 (2.48) | -2.0 (2.17)
  Change at week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 12 | -1.7 (2.20) |  |  | -3.3 (2.53) | -2.5 (2.58)
  Change at week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 20 |  | -3.1 (2.55) | -2.6 (2.76) | -4.0 (3.09) | -3.8 (2.68)
  Change at week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 24 |  | -3.7 (2.35) | -3.0 (3.15) | -4.5 (2.88) | -4.6 (2.71)
  Change at week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 28 |  | -3.8 (2.69) | -3.9 (3.22) | -4.6 (2.89) | -5.2 (2.79)
  Change at week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 32 |  | -3.9 (2.68) | -4.5 (3.28) | -4.7 (3.07) | -5.6 (3.11)
  Change at week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 36 |  | -4.8 (3.14) | -4.7 (3.39) | -4.9 (2.89) | -5.8 (3.18)
  Change at week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 40 |  | -5.0 (3.35) | -5.3 (3.12) | -5.1 (3.10) | -5.9 (3.01)
  Change at week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 44 |  | -5.0 (3.55) | -5.5 (2.89) | -5.2 (3.30) | -5.9 (3.14)
  Change at week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 48 |  | -5.3 (3.58) | -5.5 (2.90) | -5.3 (3.20) | -6.3 (3.17)
  Change at week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 52 |  | -5.6 (3.51) | -5.6 (3.00) | -5.7 (3.12) | -6.6 (3.17)
  Change at week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 60 |  | -5.5 (3.19) | -6.0 (3.06) | -5.6 (3.18) | -6.9 (3.25)
  Change at week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Change at week 72 |  | -6.5 (2.64) | -6.6 (2.65) | -6.3 (2.59) | -7.7 (2.78)
  Change at week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Change at week 84 |  | -7.5 (2.80) | -6.6 (3.45) | -6.0 (2.89) | -8.0 (2.79)

6. Secondary Outcome: Percentage of Participants Who Achieved a PPPASI-50 Response
Description: PPPASI assesses severity of PPP lesions and their response to therapy. In PPPASI system, palms and soles are divided into 4 regions: right palm, left palm, right sole, and left sole, that account for 20%, 20%, 30%, and 30%, respectively, of TSA of palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicles, and desquamation/scales, each rated on a scale of 0 to 4. PPPASI produces a score range from 0 to 72. Higher score indicates more severe disease. PPPASI-50 response represents participants who achieved at least a 50% improvement from baseline in the PPPASI score. Participants were analyzed according to the treatment at Week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 1.9 |  |  | 3.7 | 1.9
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 5.7 |  |  | 9.3 | 11.5
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 11.3 |  |  | 29.6 | 25.0
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 26.4 |  |  | 48.1 | 30.8
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 52.0 | 42.3 | 64.8 | 51.9
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 56.0 | 42.3 | 79.6 | 59.6
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 56.0 | 65.4 | 74.1 | 75.0
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 68.0 | 61.5 | 74.1 | 73.1
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 64.4 | 73.1 | 81.5 | 75.0
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 68.0 | 76.9 | 81.5 | 80.8
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 64.0 | 76.9 | 79.6 | 76.9
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 68.0 | 84.6 | 83.3 | 80.8
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 76.0 | 73.1 | 83.3 | 84.6
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 80.0 | 80.8 | 79.6 | 84.6
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 90.5 | 83.3 | 88.9 | 93.2
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 85.7 | 87.5 | 88.9 | 95.3

7. Secondary Outcome: Percentage of Participants Who Achieved a PPPASI-75 Response
Description: PPPASI assesses severity of PPP lesions and their response to therapy. In PPPASI system, palms and soles are divided into 4 regions: right palm, left palm, right sole, and left sole, that account for 20%, 20%, 30%, and 30%, respectively, of TSA of palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicles, and desquamation/scales, each rated on a scale of 0 to 4. PPPASI produces a score range from 0 to 72. Higher score indicates more severe disease. PPPASI-75 response represents participants who achieved at least a 75% improvement from baseline in the PPPASI score. Participants were analyzed according to the treatment at Week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as nonresponders at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 1.9 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 1.9 | 1.9
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 1.9 |  |  | 5.6 | 3.8
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 13 | 11.5
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 3.8 |  |  | 20.4 | 11.5
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 8.0 | 3.8 | 24.1 | 13.5
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 8.0 | 3.8 | 27.8 | 26.9
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 8.0 | 23.1 | 42.6 | 36.5
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 24.0 | 30.0 | 48.1 | 48.1
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 36.0 | 38.5 | 48.1 | 55.8
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 44.0 | 46.2 | 44.4 | 57.7
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 40.0 | 50.0 | 50.0 | 57.7
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 48.0 | 50.0 | 51.9 | 59.6
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 44.0 | 46.2 | 55.6 | 59.6
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 40.0 | 50.0 | 63.0 | 69.2
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 52.4 | 66.7 | 73.3 | 72.7
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 61.9 | 66.7 | 68.9 | 81.4

8. Secondary Outcome: Percentage of Participants Who Achieved a PPPASI-90 Response
Description: PPPASI assesses severity of PPP lesions and their response to therapy. In PPPASI system, palms and soles are divided into 4 regions: right palm, left palm, right sole, and left sole, that account for 20%, 20%, 30%, and 30%, respectively, of TSA of palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicles, and desquamation/scales, each rated on a scale of 0 to 4. PPPASI produces a score range from 0 to 72. Higher score indicates more severe disease. PPPASI-90 response represents participants who achieved at least a 90% improvement from baseline in the PPPASI score. Participants were analyzed according to the treatment at Week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 1.9 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 1.9 | 0
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 1.9
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 1.9 | 3.8
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 0 |  |  | 1.9 | 3.8
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 0 | 0 | 5.6 | 7.7
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 0 | 0 | 9.3 | 9.6
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 0 | 0 | 11.1 | 11.5
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 0 | 11.5 | 14.8 | 19.2
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 8.0 | 11.5 | 16.7 | 15.4
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 16.0 | 15.4 | 16.7 | 17.3
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 20.0 | 15.4 | 20.4 | 17.3
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 28.0 | 26.9 | 24.1 | 28.8
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 32.0 | 23.1 | 29.6 | 36.5
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 20.0 | 34.6 | 35.2 | 44.2
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 28.6 | 29.2 | 37.8 | 52.3
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 47.6 | 41.7 | 31.1 | 51.2

9. Secondary Outcome: Percentage of Participants Who Achieved a PPPASI-100 Response
Description: PPPASI assesses severity of PPP lesions and their response to therapy. In PPPASI system, palms and soles are divided into 4 regions: right palm, left palm, right sole, and left sole, that account for 20%, 20%, 30%, and 30%, respectively, of TSA of palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicles, and desquamation/scales, each rated on a scale of 0 to 4. PPPASI produces a score range from 0 to 72. Higher score indicates more severe disease. PPPASI-100 response represents participants who achieved at least a 100% improvement from baseline in the PPPASI score. Participants were analyzed according to the treatment at Week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 0 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 0 | 0
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 0
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 0 | 1.9
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 0 |  |  | 0 | 1.9
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 0 | 0 | 0 | 3.8
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 0 | 0 | 0 | 1.9
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 0 | 0 | 0 | 1.9
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 0 | 0 | 0 | 1.9
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 4.0 | 0 | 0 | 1.9
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 4.0 | 0 | 1.9 | 1.9
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 4.0 | 3.8 | 7.4 | 1.9
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 4.0 | 3.8 | 9.3 | 3.8
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 4.8 | 0 | 8.9 | 11.4
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 4.8 | 0 | 2.2 | 14.0

10. Secondary Outcome: Percentage of Participants Who Achieved a PPSI-50 Response
Description: as for outcome 2
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 1.9 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 9.3 | 5.8
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 24.1 | 3.8
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 7.5 |  |  | 27.8 | 15.4
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 11.3 |  |  | 35.2 | 19.2
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 24.0 | 15.4 | 38.9 | 28.8
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 28.0 | 26.9 | 48.1 | 42.3
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 40.0 | 34.6 | 50.0 | 48.1
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 40.0 | 46.2 | 53.7 | 57.7
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 48.0 | 46.2 | 48.1 | 63.5
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 48.0 | 53.8 | 57.4 | 63.5
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 48.0 | 57.7 | 50.0 | 65.4
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 52.0 | 50.0 | 51.9 | 69.2
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 52.0 | 57.7 | 61.1 | 69.2
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 56.0 | 65.4 | 61.1 | 75.0
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 61.9 | 83.3 | 71.1 | 81.8
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 81.0 | 79.2 | 66.7 | 83.7

11. Secondary Outcome: Percentage of Participants Who Achieved a PPSI-75 Response
Description: as for outcome 2
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 0 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 0 | 1.9
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 1.9
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 5.6 | 5.8
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 0 |  |  | 11.1 | 1.9
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 4.0 | 0 | 14.8 | 9.6
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 0 | 0 | 16.7 | 11.5
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 0 | 11.5 | 11.1 | 17.3
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 0 | 19.2 | 16.7 | 28.8
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 16.0 | 19.2 | 20.4 | 28.8
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 28.0 | 26.9 | 22.2 | 26.9
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 32.0 | 23.1 | 31.5 | 30.8
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 32.0 | 26.9 | 33.3 | 34.6
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 36.0 | 23.1 | 33.3 | 42.3
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 20.0 | 30.8 | 37.0 | 48.1
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 33.3 | 37.5 | 40.0 | 56.8
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 57.1 | 45.8 | 33.3 | 62.8

12. Secondary Outcome: Percentage of Participants Who Achieved a PPSI-90 Response
Description: PPSI assesses the severity of PPP lesions and their response to therapy with a score ranging from 0 to 12. A higher score indicates more severe disease. In the PPSI system, the more severely affected location (palms or soles) were to be identified as the evaluation sites at screening that to be assessed at all subsequent visits. Evaluation sites were assessed separately for erythema, pustules/vesicles and desquamation/scale, for most severe skin lesion rated on a scale of 0 to 4. PPSI 90 response represents participants who achieved at least a 90% improvement from baseline in the PPSI score. Participants were analyzed according to the treatment at Week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 0 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 0 | 0
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 1.9
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 0 | 1.9
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 0 |  |  | 1.9 | 1.9
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 0 | 0 | 0 | 1.9
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 0 | 0 | 0 | 3.8
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 0 | 0 | 3.7 | 3.8
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 0 | 11.5 | 3.7 | 7.7
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 4.0 | 7.7 | 1.9 | 9.6
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 8.0 | 7.7 | 5.6 | 9.6
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 12.0 | 7.7 | 16.7 | 11.5
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 16.0 | 7.7 | 11.1 | 17.3
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 20.0 | 11.5 | 16.7 | 17.3
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 20.0 | 15.4 | 13.0 | 25.0
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 23.8 | 16.7 | 22.2 | 25.0
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 28.6 | 29.2 | 17.8 | 32.6

13. Secondary Outcome: Percentage of Participants Who Achieved a PPSI-100 Response
Description: as for outcome 2
Time Frame: Week 2, 4, 8, 12, 20, 24, 28, 32, 36, 40, 44, 48, 52, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 0 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 0 | 0
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 0
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 0 | 1.9
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 0 |  |  | 0 | 1.9
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 0 | 0 | 0 | 3.8
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 0 | 0 | 0 | 3.8
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 4.0 | 0 | 0 | 1.9
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 0 | 0 | 0 | 1.9
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 4.0 | 0 | 5.6 | 1.9
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 8.0 | 0 | 3.7 | 5.8
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 8.0 | 3.8 | 11.1 | 5.8
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 8.0 | 3.8 | 9.3 | 7.7
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 4.8 | 0 | 11.1 | 15.9
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 9.5 | 4.2 | 6.7 | 20.9

14. Secondary Outcome: Percentage of Participants in Each Categories of Physician's Global Assessment (PGA) Score
Description: The PGA documents the Physician's Global Assessment of the PPP overall skin lesions status. The participant's PPP is assessed as clear (0), almost clear (1), mild (2), moderate (3), severe (4), or very severe (5). Participants were analyzed according to the treatment at week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders at week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: Clear (0): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2: Clear (0) | 0 |  |  | 0 | 0
  Week 2: Almost clear (1): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2: Almost clear (1) | 0 |  |  | 0 | 0
  Week 2: Mild (2): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2: Mild (2) | 5.7 |  |  | 1.9 | 7.7
  Week 2: Moderate (3): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2: Moderate (3) | 39.6 |  |  | 46.3 | 44.2
  Week 2: Severe (4): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2: Severe (4) | 47.2 |  |  | 48.1 | 36.5
  Week 2: Very severe (5): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2: Very severe (5) | 7.5 |  |  | 3.7 | 11.5
  Week 4: Clear (0): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4: Clear (0) | 0 |  |  | 0 | 0
  Week 4: Almost clear (1): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4: Almost clear (1) | 0 |  |  | 0 | 0
  Week 4: Mild (2): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4: Mild (2) | 7.5 |  |  | 5.6 | 9.6
  Week 4: Moderate (3): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4: Moderate (3) | 39.6 |  |  | 53.7 | 38.5
  Week 4: Severe (4): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4: Severe (4) | 45.3 |  |  | 38.9 | 48.1
  Week 4: Very severe (5): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4: Very severe (5) | 7.5 |  |  | 1.9 | 3.8
  Week 8: Clear (0): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8: Clear (0) | 0 |  |  | 0 | 0
  Week 8: Almost clear (1): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8: Almost clear (1) | 0 |  |  | 0 | 1.9
  Week 8: Mild (2): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8: Mild (2) | 15.1 |  |  | 18.5 | 11.5
  Week 8: Moderate (3): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8: Moderate (3) | 37.7 |  |  | 61.1 | 48.1
  Week 8: Severe (4): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8: Severe (4) | 41.5 |  |  | 20.4 | 36.5
  Week 8: Very severe (5): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8: Very severe (5) | 5.7 |  |  | 0 | 1.9
  Week 12: Clear (0): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12: Clear (0) | 0 |  |  | 0 | 1.9
  Week 12: Almost clear (1): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12: Almost clear (1) | 0 |  |  | 0 | 3.8
  Week 12: Mild (2): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12: Mild (2) | 17.0 |  |  | 31.5 | 17.3
  Week 12: Moderate (3): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12: Moderate (3) | 43.4 |  |  | 48.1 | 44.2
  Week 12: Severe (4): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12: Severe (4) | 32.1 |  |  | 20.4 | 30.8
  Week 12: Very severe (5): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12: Very severe (5) | 7.5 |  |  | 0 | 1.9
  Week 16: Clear (0): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16: Clear (0) | 0 |  |  | 0 | 1.9
  Week 16: Almost clear (1): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16: Almost clear (1) | 5.7 |  |  | 7.4 | 0
  Week 16: Mild (2): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16: Mild (2) | 15.1 |  |  | 38.9 | 25.0
  Week 16: Moderate (3): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16: Moderate (3) | 43.4 |  |  | 44.4 | 50.0
  Week 16: Severe (4): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16: Severe (4) | 28.3 |  |  | 9.3 | 19.2
  Week 16: Very severe (5): number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16: Very severe (5) | 7.5 |  |  | 0 | 3.8
  Week 20: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20: Clear (0) |  | 0 | 0 | 0 | 0
  Week 20: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20: Almost clear (1) |  | 8.0 | 3.8 | 9.3 | 7.7
  Week 20: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20: Mild (2) |  | 28.0 | 23.1 | 38.9 | 25.0
  Week 20: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20: Moderate (3) |  | 32.0 | 42.3 | 44.4 | 53.8
  Week 20: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20: Severe (4) |  | 28.0 | 23.1 | 7.4 | 9.6
  Week 20: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20: Very severe (5) |  | 4.0 | 7.7 | 0 | 3.8
  Week 24: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24: Clear (0) |  | 0 | 0 | 0 | 1.9
  Week 24: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24: Almost clear (1) |  | 8.0 | 3.8 | 14.8 | 13.5
  Week 24: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24: Mild (2) |  | 36.0 | 42.3 | 40.7 | 42.7
  Week 24: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24: Moderate (3) |  | 36.0 | 26.9 | 37.0 | 42.3
  Week 24: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24: Severe (4) |  | 16.0 | 23.1 | 7.4 | 7.7
  Week 24: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24: Very severe (5) |  | 4.0 | 3.8 | 0 | 1.9
  Week 28: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28: Clear (0) |  | 0 | 0 | 0 | 3.8
  Week 28: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28: Almost clear (1) |  | 8.0 | 3.8 | 14.8 | 13.5
  Week 28: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28: Mild (2) |  | 28.0 | 46.2 | 46.3 | 40.4
  Week 28: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28: Moderate (3) |  | 48.0 | 23.1 | 33.3 | 38.5
  Week 28: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28: Severe (4) |  | 12.0 | 26.9 | 5.6 | 1.9
  Week 28: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28: Very severe (5) |  | 4.0 | 0 | 0 | 1.9
  Week 32: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32: Clear (0) |  | 0 | 0 | 0 | 1.9
  Week 32: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32: Almost clear (1) |  | 8.0 | 11.5 | 16.7 | 23.1
  Week 32: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32: Mild (2) |  | 32.0 | 46.2 | 46.3 | 36.5
  Week 32: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32: Moderate (3) |  | 48.0 | 26.9 | 31.5 | 26.9
  Week 32: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32: Severe (4) |  | 12.0 | 15.4 | 5.6 | 9.6
  Week 32: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 36: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36: Clear (0) |  | 0 | 0 | 0 | 1.9
  Week 36: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36: Almost clear (1) |  | 12.0 | 19.2 | 22.2 | 23.1
  Week 36: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36: Mild (2) |  | 36.0 | 42.3 | 44.4 | 38.5
  Week 36: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36: Moderate (3) |  | 32.0 | 30.8 | 29.6 | 30.8
  Week 36: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36: Severe (4) |  | 20.0 | 7.7 | 3.7 | 3.8
  Week 36: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 40: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40: Clear (0) |  | 0 | 0 | 0 | 1.9
  Week 40: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40: Almost clear (1) |  | 20.0 | 23.1 | 24.1 | 26.9
  Week 40: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40: Mild (2) |  | 28.0 | 38.5 | 37.0 | 38.5
  Week 40: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40: Moderate (3) |  | 36.0 | 30.8 | 33.0 | 28.8
  Week 40: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40: Severe (4) |  | 16.0 | 7.7 | 5.6 | 1.9
  Week 40: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 44: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44: Clear (0) |  | 4.0 | 0 | 3.7 | 1.9
  Week 44: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44: Almost clear (1) |  | 24.0 | 15.4 | 24.1 | 32.7
  Week 44: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44: Mild (2) |  | 24.0 | 50.0 | 40.7 | 32.7
  Week 44: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44: Moderate (3) |  | 28.0 | 30.8 | 25.9 | 26.9
  Week 44: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44: Severe (4) |  | 20.0 | 3.8 | 5.6 | 3.8
  Week 44: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 48: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48: Clear (0) |  | 4.0 | 0 | 1.9 | 3.8
  Week 48: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48: Almost clear (1) |  | 32.0 | 26.9 | 29.6 | 25.0
  Week 48: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48: Mild (2) |  | 8.0 | 38.5 | 35.2 | 50.0
  Week48: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week48: Moderate (3) |  | 40.0 | 30.8 | 27.0 | 15.4
  Week 48: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48: Severe (4) |  | 16.0 | 3.8 | 5.6 | 3.8
  Week 48: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 52: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52: Clear (0) |  | 4.0 | 3.8 | 7.4 | 3.8
  Week 52: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52: Almost clear (1) |  | 28.0 | 23.1 | 24.1 | 21.2
  Week 52: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52: Mild (2) |  | 20.0 | 50.0 | 40.7 | 51.9
  Week 52: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52: Moderate (3) |  | 32.0 | 19.2 | 24.1 | 21.2
  Week 52: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52: Severe (4) |  | 16.0 | 3.8 | 3.7 | 0
  Week 52: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 60: Clear (0): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60: Clear (0) |  | 4.0 | 3.8 | 9.3 | 5.8
  Week 60: Almost clear (1): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60: Almost clear (1) |  | 20.0 | 23.1 | 25.9 | 44.2
  Week 60: Mild (2): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60: Mild (2) |  | 24.0 | 46.2 | 38.9 | 26.9
  Week 60: Moderate (3): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60: Moderate (3) |  | 40.0 | 26.9 | 20.4 | 21.2
  Week 60: Severe (4): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60: Severe (4) |  | 12.0 | 0 | 5.6 | 0
  Week 60: Very severe (5): number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60: Very severe (5) |  | 0 | 0 | 0 | 1.9
  Week 72: Clear (0): number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72: Clear (0) |  | 4.8 | 0 | 11.1 | 13.6
  Week 72: Almost clear (1): number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72: Almost clear (1) |  | 19.0 | 37.5 | 28.9 | 38.6
  Week 72: Mild (2): number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72: Mild (2) |  | 52.4 | 50.0 | 42.2 | 34.1
  Week 72: Moderate (3): number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72: Moderate (3) |  | 19.0 | 12.5 | 17.8 | 13.6
  Week 72: Severe (4): number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72: Severe (4) |  | 4.8 | 0 | 0 | 0
  Week 72: Very severe (5): number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72: Very severe (5) |  | 0 | 0 | 0 | 0
  Week 84: Clear (0): number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84: Clear (0) |  | 4.8 | 0 | 4.4 | 16.3
  Week 84: Almost clear (1): number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84: Almost clear (1) |  | 38.1 | 54.2 | 33.3 | 37.2
  Week 84: Mild (2): number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84: Mild (2) |  | 38.1 | 29.2 | 42.2 | 34.9
  Week 84: Moderate (3): number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84: Moderate (3) |  | 4.8 | 12.5 | 13.3 | 9.3
  Week 84: Severe (4): number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84: Severe (4) |  | 14.3 | 0 | 6.7 | 2.3
  Week 84: Very severe (5): number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84: Very severe (5) |  | 0 | 4.2 | 0 | 0

15. Secondary Outcome: Percentage of Participants Who Achieved a PGA Score of Cleared (0) or Almost Cleared (1)
Description: The PGA documents the Physician's Global Assessment of the participant's palmoplantar overall skin lesions status. The participant's PPP is assessed as clear (0), almost clear (1), mild (2), moderate (3), severe (4), or very severe (5). Participants who achieved a PGA score of clear (0) or almost clear (1) were reported. Participants were analyzed according to the treatment at week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders through Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 0 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 0 | 0
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 1.9
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 0 | 5.8
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 5.7 |  |  | 7.4 | 1.9
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 8.0 | 3.8 | 9.3 | 7.7
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 8.0 | 3.8 | 14.8 | 15.4
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 8.0 | 3.8 | 14.8 | 17.3
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 8.0 | 11.5 | 16.7 | 25.0
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 12.0 | 19.2 | 22.2 | 25.0
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 20.0 | 23.1 | 24.1 | 28.8
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 28.0 | 15.4 | 27.8 | 34.6
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 36.0 | 26.9 | 31.5 | 28.8
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 32.0 | 26.9 | 31.5 | 25.0
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 24.0 | 26.9 | 35.2 | 50.0
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 23.8 | 37.5 | 40.0 | 52.3
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 42.9 | 54.2 | 37.8 | 53.5

16. Secondary Outcome: Percentage of Participants Who Achieved a PGA Score of Cleared (0) or Almost Cleared (1) and Had at Least a 2-Grade Improvement
Description: The PGA documents the Physician's Global Assessment of the participant's palmoplantar overall skin lesions status. The participant's PPP is assessed as clear (0), almost clear (1), mild (2), moderate (3), severe (4), or very severe (5). Participants who achieved a PGA score of clear (0) or almost clear (1) and had at least a 2-grade improvement from baseline were reported. Participants were analyzed according to the treatment at week 0 or 16. Participants who discontinue study agent as they met a TF criterion were considered as non-responders through Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72 and Week 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Percentage of participants
  Week 2: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 2 | 0 |  |  | 0 | 0
  Week 4: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 4 | 0 |  |  | 0 | 0
  Week 8: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 8 | 0 |  |  | 0 | 1.9
  Week 12: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 12 | 0 |  |  | 0 | 5.8
  Week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Week 16 | 5.7 |  |  | 7.4 | 1.9
  Week 20: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 20 |  | 8.0 | 3.8 | 9.3 | 7.7
  Week 24: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 24 |  | 8.0 | 3.8 | 14.8 | 15.4
  Week 28: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 28 |  | 8.0 | 3.8 | 14.8 | 17.3
  Week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 32 |  | 8.0 | 11.5 | 16.7 | 25.0
  Week 36: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 36 |  | 12.0 | 19.2 | 22.2 | 25.0
  Week 40: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 40 |  | 20.0 | 23.1 | 24.1 | 28.8
  Week 44: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 44 |  | 28.0 | 15.4 | 27.8 | 34.6
  Week 48: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 48 |  | 36.0 | 26.9 | 31.5 | 28.8
  Week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 52 |  | 32.0 | 26.9 | 31.5 | 25.0
  Week 60: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Week 60 |  | 24.0 | 26.9 | 35.2 | 50.0
  Week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Week 72 |  | 23.8 | 37.5 | 40.0 | 52.3
  Week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Week 84 |  | 42.9 | 54.2 | 37.8 | 53.5

17. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Score
Description: The DLQI is a dermatology-specific quality of life (QOL) instrument designed to assess the impact of the disease on a participant's QOL. It is a 10-item participant-reported outcome questionnaire that, in addition to evaluating overall QOL, can be used to assess 6 different aspects that may affect QOL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The DLQI produces a numeric score that can range from 0 to 30. Higher score indicates more severe disease. Participants were analyzed according to the treatment at week 0 or 16. Participants who discontinue study agent as they met a TF criterion, their baseline value carried forward to the post-baseline attending visits before and at Week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Baseline, Week 16, 32, 52, 72 and Week 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Units on a scale
  Change at week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 16 | -1.8 (4.71) |  |  | -5.0 (5.59) | -3.1 (3.49)
  Change at week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 32 |  | -4.3 (5.25) | -4.2 (5.09) | -5.2 (5.90) | -4.2 (4.18)
  Change at week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 52 |  | -4.8 (5.74) | -5.2 (5.10) | -5.7 (6.05) | -4.9 (5.24)
  Change at week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Change at week 72 |  | -5.5 (5.82) | -5.8 (4.28) | -6.2 (5.78) | -5.8 (5.20)
  Change at week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Change at week 84 |  | -6.0 (5.29) | -5.6 (4.66) | -6.4 (5.59) | -6.3 (5.41)

18. Secondary Outcome: Change From Baseline in the 36-Item Short-Form Health Assessment Questionnaire (SF-36) Physical Component Summary (PCS) Score
Description: SF-36 consists of 8 individual domains, which are weighted sums of questions in their section. 8 domains are: vitality(VT), physical functioning(PF), bodily pain(BP), general health(GH), Role-Physical(RP), Role-Emotional(RE), social functioning(SF) and mental health(MH). Each of these 8 scales (domains) is scored from 0 to 100 with higher scores indicating better health. Based on scale scores, summary PCS is derived. Scales contributing most to the scoring of the SF-36 PCS include PF,RP,BP and GH. Other domains not noted contribute to scoring but to a lesser degree. Scoring is derived based on an algorithm as presented in Japanese edition manual. Summary PCS score is also scaled from 0 to 100 with higher scores indicating better health. Participants who discontinue study agent as they met a TF criterion, their baseline value carried forward to post-baseline attending visits before and at week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Baseline, Week 16, 32, 52, 72 and Week 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Units on a scale
  Change at week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 16 | 1.27 (9.177) |  |  | 4.67 (13.753) | 3.34 (10.259)
  Change at week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 32 |  | 5.46 (16.226) | 7.16 (11.507) | 8.31 (15.510) | 4.82 (9.975)
  Change at week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 52 |  | 7.92 (14.580) | 8.18 (11.320) | 7.35 (17.320) | 6.47 (11.466)
  Change at week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Change at week 72 |  | 9.02 (17.049) | 7.02 (11.806) | 6.75 (15.098) | 7.55 (11.453)
  Change at week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Change at week 84 |  | 9.29 (19.175) | 9.01 (12.964) | 7.06 (15.034) | 6.75 (13.619)

19. Secondary Outcome: Change From Baseline in the 36-Item Short-Form Health Assessment Questionnaire (SF-36) Mental Component Summary (MCS) Score
Description: as for outcome 18
Time Frame: Baseline, Week 16, 32, 52, 72 and Week 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Units on a scale
  Change at week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 16 | 1.20 (7.823) |  |  | 0.64 (7.880) | 0.66 (7.055)
  Change at week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 32 |  | 2.19 (10.277) | 1.10 (7.579) | 0.52 (8.124) | 0.59 (7.639)
  Change at week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 52 |  | 1.44 (9.980) | 0.39 (7.431) | 1.69 (7.866) | 0.69 (7.354)
  Change at week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Change at week 72 |  | 1.51 (10.679) | 0.02 (8.686) | 2.19 (7.112) | 0.92 (6.797)
  Change at week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Change at week 84 |  | 1.72 (8.740) | 0.78 (6.975) | 2.51 (8.428) | 2.58 (7.977)

20. Secondary Outcome: Change From Baseline in the EuroQOL-5 Dimensions Questionnaire Visual Analogue Scale (EQ-5D VAS) Score
Description: EQ-5D is designed for self-completion by participants and consists of EQ-5D descriptive system and the EQ visual analog scale (EQ VAS). The EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and unable. The EQ VAS records the respondent's self-rated health on a vertical, VAS where the endpoints are labeled 'Best imaginable health state' (score of 100) and 'Worst imaginable health state' (score of 0). Participants were analyzed according to the treatment at week 0 or 16. Participants who discontinue study agent as they met a TF criterion their baseline value carried forward to the post-baseline attending visits before and at week 16 and after TF were applied, remaining missing data were handled with LOCF till Week 60.
Time Frame: Baseline, Week 16, 32, 52, 72 and Week 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
Number analyzed (Participants) | 53 | 25 | 26 | 54 | 52
Units on a scale
  Change at week 16: number analyzed (Participants) | 53 | 0 | 0 | 54 | 52
  Change at week 16 | -0.1 (14.33) |  |  | 8.3 (21.25) | 8.5 (15.59)
  Change at week 32: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 32 |  | 8.0 (25.36) | 6.5 (15.75) | 10.2 (21.88) | 5.9 (15.98)
  Change at week 52: number analyzed (Participants) | 0 | 25 | 26 | 54 | 52
  Change at week 52 |  | 13.0 (24.69) | 5.6 (16.28) | 13.9 (22.19) | 7.9 (15.19)
  Change at week 72: number analyzed (Participants) | 0 | 21 | 24 | 45 | 44
  Change at week 72 |  | 13.0 (21.59) | 8.7 (21.08) | 12.9 (22.43) | 10.5 (17.11)
  Change at week 84: number analyzed (Participants) | 0 | 21 | 24 | 45 | 43
  Change at week 84 |  | 6.7 (24.71) | 10.0 (19.55) | 10.5 (21.53) | 8.7 (18.42)

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) up to Week 84
Arm/Group | Placebo | Placebo Then Guselkumab 100 mg | Placebo Then Guselkumab 200 mg | Guselkumab 100 mg | Guselkumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/25 | 0/26 | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/53 | 3/25 | 1/26 | 3/54 | 5/52
Other Adverse Events (participants affected / at risk) | 34/53 | 23/25 | 22/26 | 44/54 | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Placebo Then Guselkumab 100 mg (N=25) | Placebo Then Guselkumab 200 mg (N=26) | Guselkumab 100 mg (N=54) | Guselkumab 200 mg (N=52)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Heat Stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Synovial Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung Carcinoma Cell Type Unspecified Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Abortion Induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Medical Device Removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=53) | Placebo Then Guselkumab 100 mg (N=25) | Placebo Then Guselkumab 200 mg (N=26) | Guselkumab 100 mg (N=54) | Guselkumab 200 mg (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1
Corneal Perforation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Dental Caries (Gastrointestinal disorders) | 2 | 2 | 3 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 2
Injection Site Erythema (General disorders) | 0 | 3 | 5 | 4 | 10
Injection Site Induration (General disorders) | 0 | 1 | 1 | 1 | 1
Injection Site Pruritus (General disorders) | 1 | 2 | 3 | 1 | 5
Injection Site Swelling (General disorders) | 0 | 0 | 3 | 2 | 3
Malaise (General disorders) | 1 | 1 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 2 | 2 | 3 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 3
Gingivitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 9 | 17 | 14 | 20 | 25
Oral Herpes (Infections and infestations) | 2 | 0 | 3 | 0 | 3
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Tinea Pedis (Infections and infestations) | 2 | 0 | 0 | 5 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Vaginal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2
Ligament Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Traumatic Ulcer (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Peripheral Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic Pigmented Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 6 | 8
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 4
Eczema Nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Polymorphic Light Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3
Skin Discomfort (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 7
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 1
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0/24 | 0 | 2
Oral Lichen Planus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0/24 | 1 | 2/42
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Helicobacter Gastritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Infected Dermal Cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Myringitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 2 | 1 | 2
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02641730/Prot_001.pdf
  • Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT02641730/SAP_000.pdf